CLINICAL TRIAL: NCT04175132
Title: Interventional, Open-label, Positron Emission Tomography (PET) Study With [11C]-PXT012253 Investigating the Brain mGlu4 Receptor Occupancy, Safety, Tolerability and Pharmacokinetics of Foliglurax in Healthy Subjects and Patients With Parkinson's Disease
Brief Title: Binding of Foliglurax to Regions in the Brain in Healthy Participants and in Patients With Parkinson's Disease (PD)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New efficacy data from another study
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18124A
Record Dates: First submitted 2019-11-12; First posted 2019-11-22 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Healthy; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — foliglurax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Experimental)
  Interventions: Drug: foliglurax
- PD patients (Experimental)
  Interventions: Drug: foliglurax

INTERVENTIONS:
Drug: foliglurax — Capsules of 20/80 mg foliglurax, orally. Single doses of 20-240 mg
  Arms: Healthy subjects
Drug: foliglurax — Capsules of 20/80 mg foliglurax, orally. Single doses of 20-160 mg
  Arms: PD patients

SUMMARY:
A study to learn how foliglurax binds in regions of the brain

DETAILED DESCRIPTION:
To study binding of foliglurax to mGlu4 receptors in human brain, up to 9 healthy subjects (Part A) and up to 8 patients with Parkinson's disease (Part B) will be injected with a liquid dose of a radiolabelled tracer that allows measurement of foliglurax binding in the brain to determine to which degree foliglurax binds to regions of the brain.

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Healthy subjects
* The subject has a normal structural MRI (sMRI) scan performed in the screening period, as judged by the investigator.
* The subject is, in the opinion of the investigator, generally healthy based on the assessment of medical history, physical examination, vital signs, body weight, ECG, and the results of the haematology, clinical chemistry, urinalysis, serology, and other laboratory tests.
* The subject can tolerate confined spaces for prolonged periods of time.
* The subject is suitable for radial and/or brachial artery blood sampling and cannulation.

Part B:

* Patients with Parkinson's disease
* The subject has a normal sMRI scan performed in the screening period, as judged by the investigator.
* The patient is, in the opinion of the investigator, fit for enrolment in the study based on the assessment of medical history, physical examination, vital signs, body weight, ECG, and the results of the haematology, clinical chemistry, urinalysis, serology, and other laboratory tests.
* The patient has been diagnosed with idiopathic Parkinson's disease for ≥3 years, with a current disease severity of 2 to 4 on the modified Hoehn and Yahr scale in the OFF state.
* The patient has dyskinesia that is not too severe to cause discomfort for the patient during PET imaging and predictable OFF time
* In addition to the above criteria, the patient must, in the opinion of the investigator, also be suitable for the study and the included PET imaging sessions.
* The patient has been receiving a stable regimen of levodopa-containing therapy (total levodopa dose ≤1600 mg per day) (≥3 doses per day of standard levodopa or ≥3 doses per day of carbidopa and levodopa, sustained-release tablets or extended-release capsules of carbidopa and levodopa or benserazide and levodopa), and be on a stable regimen of permitted anti-Parkinsonian drugs (peripheral decarboxylase inhibitors, dopamine agonists [except apomorphine], monoamine oxidase type B [MAO-B] inhibitors [except safinamide], or catechol-O-methyl transferase [COMT] inhibitors) for ≥4 weeks prior to foliglurax dosing
* The patient can tolerate confined spaces for prolonged periods of time
* The patient is suitable for radial and/or brachial artery blood sampling and cannulation

Exclusion Criteria:

* The subject has any concurrent disorder that may affect the particular target or absorption, distribution, or elimination of the IMP

Other inclusion and exclusion criteria may apply.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Receptor Occupancy (RO) on the metabotropic glutamate receptor 4 (mGlu4) | From Day 1 up to Day 3
  in Healthy Participants and in Patients With Parkinson's Disease
C(PET) foliglurax | From Day 1 up to Day 3
  mean plasma concentration of foliglurax during PET measurement in Healthy Participants and in Patients With Parkinson's Disease

SECONDARY OUTCOMES:
AUC(0-24) foliglurax | From Day 1 up to Day 3
  Area under the plasma concentration curve from zero to 24 hours
Cmax foliglurax | From Day 1 up to Day 3
  Maximum observed plasma concentration of foliglurax
Tmax foliglurax | From Day 1 up to Day 3
  Corresponding time (tmax) in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Karolinska Institutet, Stockholm, Sweden